CLINICAL TRIAL: NCT00177281
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of S-CKD602 in Patients With Advanced Malignancies
Brief Title: Safety Study of S-CKD602 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: ALZA (Industry)
Responsible Party: Principal Investigator, Laura A. Pollice, Clinical Research Manager, University of Pittsburgh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-052
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: S CKD602

SUMMARY:
The purpose of this research study is to evaluate a new anti-cancer drug called S CKD602, developed by ALZA Corporation. The drug is investigational and not approved by the Food and Drug administration (FDA). The side effects (the way the drug acts in your body) and the effect it has on your disease will be studied.

DETAILED DESCRIPTION:
The main purposes of this study are:

To determine the maximum tolerated dose (highest dose that can safely be given to subjects) of S CKD602 when given every three weeks.

To determine the incidence and severity of toxicity (side-effects) of S CKD602 when given every three weeks.

To determine a subject's body handles the drug (pharmacokinetics) following administration of S CKD602.

In addition to the above, we would also like to analyze how the genes (material inside each cell that is responsible for cell functioning and appearance) found in a subject's blood affect how the study drug S-CKD602 is broken down in a subject's body. This process is referred to as "metabolic genotyping analyses". This evaluation is performed using a blood sample and is optional.

ELIGIBILITY:
Inclusion Criteria:

Male or female subjects with an age > 18 years Histologically or cytologically proven malignancy, unresponsive to curative surgery, radiotherapy, conventional chemotherapy or for which no conventional therapy exists. (Measurable or evaluable disease is desirable, but not required) Note: This study is restricted to patients with advanced solid tumors, subjects with hematological malignancies are excluded (including lymphoma and leukemia) ECOG Performance Status 0- 2 Adequate bone marrow function, without the support of cytokines and/or Epoetin Alpha within 5 days prior to dosing: Absolute neutrophil count (ANC) >1,500/mm3, platelet count > 100,000/mm3, Hgb > 9.0 g/dL. Adequate liver function: total bilirubin level < 2.0 mg/dL, ALT and AST < 2.0 x institutional upper limit of normal in the absence of liver metastasis, or < 4.0 x institutional upper limit of normal in the presence of liver metastasis.

Adequate renal function: serum creatinine < 1.5 mg/dL. At least 3 weeks since prior chemotherapy or cancer surgery (6 weeks for nitrosourea or mitomycin C).

Normal cardiac function with no history of uncontrolled heart disease. Women subjects (if of child bearing potential and sexually active) and male subjects (if sexually active with a partner of child bearing potential) must use medically acceptable methods of birth control prior to study entry and for the duration of the study. Medically acceptable methods of contraception that may be used by the subject and/or his/her partner include abstinence, birth control pills or patches, diaphragm and spermicide, IUD, condom and vaginal spermicide, surgical sterilization, post menopausal, vasectomy, and progestin implant or injection.

Written informed consent.

Exclusion Criteria:

Subject is pregnant or is breast feeding. Subject's life expectancy is less than 3 months. Subject exhibits confusion, disorientation, or has a history of major Psychiatric illness, which may potentially impair subject's understanding of the informed consent.

Subject has signs and symptoms of acute infection requiring systemic therapy. Subject has used another investigational agent within 30 days of dosing with S CKD602.

Subjects with known allergic reactions to camptothecin analogs, dextran sulfate or other components of S-CKD602 Symptomatic or uncontrolled brain leptomeningeal metastasis. CT scans are not required unless there is clinical suspicion of central nervous disease.

Not recovered from reversible toxicity of prior therapy. Subjects with known brain metastases because of their poor prognosis because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

Concurrent radiation therapy or radiation within 3 weeks of starting treatment with S-CKD602.

Concurrent anti-neoplastic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of S CKD602 when given every three weeks.
To determine the incidence and severity of toxicity of S CKD602 when given every three weeks.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of CKD 602 following administration of S CKD602.

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh K Ramanathan, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States